CLINICAL TRIAL: NCT03576716
Title: Clearance of 25-hydroxyvitamin D3 During Vitamin D3 Supplementation
Acronym: CLEAR-PLUS
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Ian deBoer, Professor, Medicine/Nephrology, University of Washington
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: STUDY00000608; R01DK099199 (NIH)
Record Dates: First submitted 2018-06-22; First posted 2018-07-03 (Actual); Results first posted 2021-09-28 (Actual); Last update posted 2022-05-17 (Actual); Status verified 2022-05

CONDITIONS: Chronic Kidney Disease
Keywords: chronic kidney disease; vitamin d catabolism
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Study Population (Experimental): D6-25-hydroxyvitamin D3 with vitamin D3
  Interventions: Drug: D6-25-hydroxyvitamin D3

INTERVENTIONS:
Drug: D6-25-hydroxyvitamin D3 — Intravenous administration of a deuterium-labeled 25(OH)D3 to evaluate the metabolic clearance of 25(OH)D3
  Other Names: stable isotope deuterium-labeled 25(OH)D3

SUMMARY:
The goal of this study is to determine how 25(OH)D3 clearance is affected by vitamin D3 supplementation using a gold standard pharmacokinetic approach.

DETAILED DESCRIPTION:
We expect that this study will enhance interpretation of available diagnostic tests, inform the results of ongoing large clinical trials of vitamin D supplements, and help develop new strategies to target vitamin D to improve health.

ELIGIBILITY:
Inclusion Criteria:

* Successful prior completion of related protocol CLEAR (NCT02937350) or CLEAR-CF (NCT03104855)
* Age ≥ 18 years
* Self-reported race Caucasian, African American, or African

Exclusion Criteria:

* Primary hyperparathyroidism
* Gastric bypass
* Tuberculosis or sarcoidosis
* Current pregnancy
* Child-Pugh Class B or C cirrhosis (i.e. cirrhosis with ascites, hepatic encephalopathy, bilirubin >=2 mg/dL, serum albumin <=3.5 g/dL, or PT >= 4 seconds)
* History of kidney transplantation (unless failed transplant now treated with hemodialysis)
* Use of 1,25(OH)2D3 or an analogue, calcimimetics, or medications known to induce CYP24A1 within 4 weeks (wash-out allowed)
* Serum calcium > 10.1 mg/dL
* Hemoglobin < 10 g/dL

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2019-07-08 (Actual); Study Completion 2021-01-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ian de Boer, MD, MS, Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No
Coded individual participant data may be shared with other researchers under mutually agreeable terms.

REFERENCES:
- [Derived] Hsu S, Zelnick LR, Lin YS, Best CM, Kestenbaum B, Thummel KE, Rose LM, Hoofnagle AN, de Boer IH. Differences in 25-Hydroxyvitamin D Clearance by eGFR and Race: A Pharmacokinetic Study. J Am Soc Nephrol. 2021 Jan;32(1):188-198. doi: 10.1681/ASN.2020050625. Epub 2020 Oct 28. PMID 33115916

RESULTS

PARTICIPANT FLOW:
Groups:
- Healthy Controls: Healthy controls defined as normal eGFR (>60 ml/min per 1.73m2)
- CKD Group: CKD group defined as those with eGFR (<60 ml/min per 1.73 m2)
Period: Overall Study
Arm/Group | Healthy Controls | CKD Group
Started | 10 | 9
Completed | 10 | 8
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Healthy Controls: Healthy Controls (n = 10)
- CKD Group: CKD Group (n = 8)
- Total: Total of all reporting groups
Arm/Group | Healthy Controls | CKD Group | Total
Number analyzed (Participants) | 10 | 8 | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 60 (6) | 69 (7) | 64 (7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 2 | 6
  Male | 6 | 6 | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 4 | 10
  White | 4 | 4 | 8
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Clearance after supplement [Mean (Standard Deviation); unit: ml/d] | 436 (135) | 322 (88) | 385 (128)

OUTCOME MEASURES:

1. Primary Outcome: Change in Metabolic Clearance of D6-25(OH)D3
Description: Metabolic clearance is calculated as the administered dose of 25(OH)D3 divided by the area under the plasma concentration-time curve (AUC). AUC is calculated using the linear trapezoidal method. Change in clearance of D6-25(OH)D3 will be calculated as D6-25(OH)D3 clearance measured during CLEAR-PLUS minus D6-25(OH)D3 clearance previously measured during participation in the related study protocol (without vitamin D3 supplementation). Concentration was measured at 5 minutes, 4 hours, and at 1, 4, 7, 14, 21, 28, 42, and 56 days post administration. The change listed is between two timepoints.
Time Frame: Baseline, 6 months
Measure: Mean (95% Confidence Interval); unit: ml/d
Groups:
- CKD Group: CKD group defined as those with eGFR (<60ml/min per 1.73m2)
Arm/Group | Healthy Controls | CKD Group
Number analyzed (Participants) | 10 | 8
ml/d | 21 [-63 to 105] | 5 [-45 to 55]

2. Secondary Outcome: Change in AUC of D6-25(OH)D3
Description: AUC is calculated using the linear trapezoidal method. Change in the AUC of D6-25(OH)D3 will be calculated as D6-25(OH)D3 AUC measured during CLEAR-PLUS minus D6-25(OH)D3 AUC previously measured during participation in the related study protocol (without vitamin D3 supplementation). Concentration was measured at 5 minutes, 4 hours, and at 1, 4, 7, 14, 21, 28, 42, and 56 days post administration. The change listed is between two timepoints.
Time Frame: Baseline, 6 months
Measure: Mean (Standard Deviation); unit: ng x day/mL
Groups:
- Healthy Controls: Healthy controls defined as normal eGFR (>60ml/min per 1.73m2)
Arm/Group | Healthy Controls | CKD Group
Number analyzed (Participants) | 10 | 8
ng x day/mL | 0.07 (11.2) | -2.58 (7.51)

3. Secondary Outcome: Change in Terminal Half-life of D6-25(OH)D3
Description: Terminal half-life is equal to ln2/k, where k is the slope of the terminal regression line estimated using ≥3 plasma concentrations. Change in the terminal half-life of D6-25(OH)D3 will be calculated as D6-25(OH)D3 half-life measured during CLEAR-PLUS minus D6-25(OH)D3 half-life previously measured during participation in the related study protocol (without vitamin D3 supplementation). Concentration was measured at 5 minutes, 4 hours, and at 1, 4, 7, 14, 21, 28, 42, and 56 days post administration. The change listed is between two timepoints.
Time Frame: Baseline, 6 months
Measure: Mean (95% Confidence Interval); unit: d
Arm/Group | Healthy Controls | CKD Group
Number analyzed (Participants) | 10 | 8
d | -1.3 [-6.3 to 3.8] | 1.2 [-5.1 to 7.4]

4. Secondary Outcome: Change in Volume of Distribution of D6-25(OH)D3
Description: Volume of distribution in the central compartment is calculated as dose/C0, where dose is the administered dose of 25(OH)D3 and C0 is the initial (estimated) concentration of drug in plasma. Change in the volume of distribution of D6-25(OH)D3 will be calculated as D6-25(OH)D3 volume of distribution measured during CLEAR-PLUS minus D6-25(OH)D3 volume of distribution previously measured during participation in the related study protocol (without vitamin D3 supplementation). Concentration was measured at 5 minutes, 4 hours, and at 1, 4, 7, 14, 21, 28, 42, and 56 days post administration. The change listed is between two timepoints.
Time Frame: Baseline, 6 months
Measure: Mean (Standard Deviation); unit: L
Arm/Group | Healthy Controls | CKD Group
Number analyzed (Participants) | 18 | 8
L | 0.28 (4.13) | 0.55 (0.94)

5. Other Pre Specified Outcome: Changes in Metabolic Formation Clearance of D6-25(OH)D3 Metabolites.
Description: Metabolic formation clearance is calculated as the daughter metabolite plasma AUC divided by the AUC of D6-25(OH)D3 (metabolite/parent AUC ratio). AUC is calculated using the linear trapezoidal method. Changes in the metabolic formation clearance of D6-25(OH)D3 metabolites will be calculated as metabolic formation clearance measured during CLEAR-PLUS minus metabolic formation clearance previously measured during participation in the related study protocol (without vitamin D3 supplementation). Concentration was measured at 5 minutes, 4 hours, and at 1, 4, 7, 14, 21, 28, 42, and 56 days post administration. The change listed is between two timepoints.
Time Frame: Baseline, 6 months
Measure: Mean (95% Confidence Interval); unit: ratio
Arm/Group | Healthy Controls | CKD Group
Number analyzed (Participants) | 10 | 8
ratio | 0.01 [-0.03 to 0.05] | -0.02 [-0.04 to 0.002]

6. Other Pre Specified Outcome: Change in the Serum Concentration of Calcium
Description: Change in the serum concentration of calcium from baseline to 7 days after 25(OH)D3 administration. The change listed is between two timepoints.
Time Frame: Baseline, 7 days
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Healthy Controls | CKD Group
Number analyzed (Participants) | 10 | 8
mg/dl | 0.20 (0.20) | 0.28 (0.33)

7. Other Pre Specified Outcome: Change in the Serum Concentration of Creatinine
Description: Change in the serum concentration of creatinine from baseline to 7 days after 25(OH)D3 administration. The change listed is between two timepoints.
Time Frame: Baseline, 7 days
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Healthy Controls | CKD Group
Number analyzed (Participants) | 10 | 8
mg/dl | 0.03 (0.10) | -0.02 (0.15)

8. Other Pre Specified Outcome: Change in the Serum Concentration of AST
Description: Change in the serum concentration of AST from baseline to 7 days after 25(OH)D3 administration. The change listed is between two timepoints.
Time Frame: Baseline, 7 days
Measure: Mean (Standard Deviation); unit: units/L
Arm/Group | Healthy Controls | CKD Group
Number analyzed (Participants) | 10 | 8
units/L | 1.30 (4.60) | -0.13 (1.36)

9. Other Pre Specified Outcome: Change in the Serum Concentration of ALT
Description: Change in the serum concentration of ALT from baseline to 7 days after 25(OH)D3 administration. The change listed is between two timepoints.
Time Frame: Baseline, 7 days
Measure: Mean (Standard Deviation); unit: units/L
Arm/Group | Healthy Controls | CKD Group
Number analyzed (Participants) | 10 | 8
units/L | 1.56 (2.83) | 0.50 (2.98)

ADVERSE EVENTS:
Time Frame: 8 weeks
Description: Everyone had the same treatment, so it's most appropriate to summarize AEs for the whole group.
Groups:
- All Participants: All Participants (N = 18). AEs were not collected by arm but altogether.
Arm/Group | All Participants
All-Cause Mortality (participants affected / at risk) | 0/18
Serious Adverse Events (participants affected / at risk) | 0/18
Other Adverse Events (participants affected / at risk) | 6/18
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | All Participants (N=18)
Sensation in arm during infusion (General disorders) | 5
Diverticulitis (Infections and infestations) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-05-18): https://cdn.clinicaltrials.gov/large-docs/16/NCT03576716/Prot_SAP_000.pdf